CLINICAL TRIAL: NCT01849549
Title: Anatomical Clinical Correlations. Neuropsychological and Brain Medical Imaging Study in Brain Damaged Subjects.
Brief Title: Neuropsychological and Brain Medical Imaging Study in Patients With Brain Damage
Acronym: CORAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012/191/HP; 2012-A01332-41 (Other: Agence Nationale de sécurité du médicament et des produits de Santé)
Record Dates: First submitted 2013-04-30; First posted 2013-05-08 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Cerebrovascular Disorders; Brain Lesions; Degenerative Diseases; Developmental Pathology
Keywords: neuropsychological Study; brain Imaging
MeSH Terms: conditions — Cerebrovascular Disorders | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- brain damaged subjects (Experimental): patients with circumscribed brain injury, selective disorders of cognitive development or degenerative disorders responsible for focal troubles
  Interventions: Behavioral: Neuropsychological testing; Other: MRI
- healthy volunteers (Sham Comparator): healthy controls
  Interventions: Behavioral: Neuropsychological testing; Other: MRI

INTERVENTIONS:
Behavioral: Neuropsychological testing — Experimental test about cognitive deficit of interest and standard neuropsychological tests.
Other: MRI — Anatomical, diffusion, and/or functional MRI

SUMMARY:
Two groups of subjects will be constitute: (i) patients with circumscribed brain injury (including stroke, vascular malformations, tumor or circumscribed infectious lesions) or degenerative disorders and selective cognitive disorders; (ii) healthy control subjects.

The objective of this project is to evaluate specific neuropsychological deficits and apply current brain imaging techniques (anatomical, diffusion, functional) to patients suffering from these cognitive deficits due to brain damage, in order to elucidate the brain mechanisms underlying these deficits.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years
* french language
* effective contraception for women during the study
* informed consent
* no alcohol intake the day before the exam
* for patients only, focal cerebral lesion (stroke, malformation, tumor, inflammatory, infectious, traumatic), neonatal pathology or degenerative disease with cognitive deficit

Exclusion Criteria:

* for healthy volunteers: previous neurological history (except non complicated migraine), previous psychiatric history (except depression with good evolution or anxiety with maximum one anxiolytic treatment), or severe cranial traumatism
* for patients: vigilance disorders, severe depression or anxiety.
* for both: psychotropic medication other than a hypnotic or an anxiolytic at low doses without dose modification for at least one month, severe visual or auditory impairment, patient without judicial or administrative liberty, measure of legal protection or no capable to express their consent, pregnancy or breastfeeding, contraindication for MRI, participation in another trial or former involvement in another trial within one month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Cognitive deficit | 3 to 6 months
  The cognitive deficit of interest will depend on the localization of the brain lesion. The outcome measure could be a standardized neuropsychological test or an experimental test specifically elaborated for this protocol.

CONTACTS AND LOCATIONS:
Overall Officials: David Wallon, Doctor, Principal Investigator — Neurology Department
Locations (1):
- CHU - Hôpitaux de Rouen, Rouen, France